CLINICAL TRIAL: NCT03873883
Title: Phase I/Ib First-in-Human Study of EOS100850 (Inupadenant) As a Single Agent and in Combination with Pembrolizumab And/or Chemotherapy in Participants with Advanced Cancers
Brief Title: First-in-Human Study of EOS100850 (Inupadenant) in Patients with Cancer
Acronym: IO-001
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: iTeos Therapeutics (Industry)
Collaborators: iTeos Belgium SA (Industry); Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: IO-001; 2018-003173-10 (EudraCT Number); Keynote A45 (Other: Merck and Co.)
Record Dates: First submitted 2019-03-06; First posted 2019-03-14 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-07

CONDITIONS: Solid Tumor, Adult
Keywords: solid; tumor; advanced cancers; pharmacokinetics; safety; inupadenant; pembrolizumab; chemotherapy
MeSH Terms: conditions — Neoplasms | interventions — pembrolizumab; Drug Therapy; Carboplatin; Paclitaxel

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (6):
- 1A Dose escalation EOS100850 (Experimental): Dose Escalation- EOS100850 Monotherapy: to confirm RP2D
  Interventions: Drug: EOS100850
- 1B Dose escalation EOS100850 and Pembrolizumab (Experimental): EOS100850 and Pembrolizumab Combination Therapy: to confirm RP2D as combination
  Interventions: Drug: EOS100850; Drug: Pembrolizumab
- 2A Dose Expansion- EOS100850 (Experimental): Dose Expansion - EOS100850 Monotherapy: to explore safety, PK, PD, and antitumor activity of inupadenant as monotherapy
  Interventions: Drug: EOS100850
- 2B Dose Expansion - EOS100850 and Pembrolizumab (Experimental): Dose Expansion - EOS100850 and Pembrolizumab Combination Therapy: to explore safety, PK, PD, and antitumor activity of inupadenant in combination with pembrolizumab in melanoma and CRPC patients
  Interventions: Drug: EOS100850; Drug: Pembrolizumab
- 2D Dose expansion - EOS100850 and Chemotherapy in TNBC (Experimental): Dose expansion - EOS100850 and Chemotherapy Combination: to explore safety, PK, PD, and antitumor activity of inupadenant in combination with chemotherapy SOC carboplatin and paclitaxel in patients with TNBC
  Interventions: Drug: EOS100850; Drug: Chemotherapy
- 3 EOS100850 in BMK-H participants (Experimental): Dose expansion - EOS100850 Monotherapy : to evaluate the safety, PD, and antitumor activity of inupadenant as monotherapy at the mono-RP2D in BMK-H participants in 4 disease-specific cohorts: NSCLC; HNSCC; EC; and other forms of cancer
  Interventions: Drug: EOS100850

INTERVENTIONS:
Drug: EOS100850 — Oral administration
  Other Names: Inupadenant
Drug: Pembrolizumab — IV Infusion
  Other Names: Keytruda; MK-3475
  Arms: 1B Dose escalation EOS100850 and Pembrolizumab; 2B Dose Expansion - EOS100850 and Pembrolizumab
Drug: Chemotherapy — Standard of Care IV Infusion
  Other Names: carboplatin and paclitaxel
  Arms: 2D Dose expansion - EOS100850 and Chemotherapy in TNBC

SUMMARY:
Multicenter, open-label, dose-escalation Phase I/Ib clinical study to evaluate the safety and tolerability, the MTD/RP2D, pharmacokinetics (PK), pharmacodynamics (PD), and antitumor activity of EOS100850 (Inupadenant) as a Single Agent and in Combination with Pembrolizumab and/or Chemotherapy in Participants with Advanced Cancers.

ELIGIBILITY:
For more information regarding participation in the Trial, please refer to your physician

Inclusion Criteria:

* Women and men ≥18 years of age with Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1
* Subject with histologically or cytologically confirmed advanced solid tumor for whom no standard treatment is further available.
* At least 4 weeks since any previous treatment for cancer
* Subject must consent to pretreatment and on treatment tumor biopsies
* Adequate organ and marrow function

Exclusion Criteria:

* Patients with primary brain tumors or primary tumors with central nervous system metastases as only location of disease. Controlled brain metastases are permitted
* Participants with second/other active cancers requiring current treatment
* Uncontrolled/significant heart disease
* Known History of chronic hepatitis, Positive test for Hepatitis B virus surface antigen or Hepatitis C antibody (except participants with liver cancer) or Human Immunodeficiency Virus/Acquired Immunodeficiency Syndrome(HIV/AIDS)
* Active/uncontrolled autoimmune disease
* Active infection

Other protocol defined inclusion/exclusion criteria could apply

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 119 (Actual)
Dates: Start 2019-02-05 (Actual); Primary Completion 2024-05-28 (Actual); Study Completion 2024-05-28 (Actual)

PRIMARY OUTCOMES:
Incidence of Dose-Limiting Toxicities (DLTs) in patients with advanced solid tumors receiving EOS100850 | During the DLT evaluation period that is cycle 1 (each cycle is 3 or 4 weeks)
  To define the maximum tolerated dose (MTD) or the recommended Phase 2 dose (RP2D) of EOS100850 in patients receiving EOS100850
Incidence and severity of AEs in patients receiving EOS100850 | Up to 30 months
  To assess safety and tolerability as measured by incidence and severity of AEs

SECONDARY OUTCOMES:
Plasma concentration of EOS100850 vs. time profiles | Up to 30 months
  Determined by inspection of the concentration-time profile
Maximum observed serum concentration (Cmax) | Up to 30 months
  Determined by inspection of the concentration-time profile
Time of maximum observed concentration (Tmax) | Up to 30 months
  Determined by inspection of the concentration-time profile
Area under the concentration-time curve in 1 dosing interval [AUC(TAU)] | Up to 30 months
  Determined by inspection of the concentration-time profile
Plasma concentration half-life (T-HALF) | Up to 30 months
  Determined by inspection of the concentration-time profile
Overall response rate per Response Evaluation Criteria In Solid Tumors (RECIST) v1.1 | Up to 30 months
  Assessment of preliminary efficacy of EOS100850

CONTACTS AND LOCATIONS:
Overall Officials: Iteos Clinical Trials, Study Director — iTeos Belgium SA
Locations (19):
- United States (3):
  - Karmanos Cancer Institute, Michigan Center, Michigan
  - John Theurer Cancer Center, Hackensack University Medical Center, Hackensack, New Jersey
  - University of Texas Health Science Center at San Antonio, San Antonio, Texas
- Belgium (4):
  - Hospital GZA Sint-Augustinus, Wilrijk, Antwerpen
  - Institut Jules Bordet, Anderlecht, Brussels Capital
  - UCL Saint-Luc, Brussels, Brussels Capital
  - UZ Ghent, Ghent, East-Flanders
- France (4):
  - Centre de Lutte Contre le Cancer (CLCC) - Universite de Lyon - Centre Leon-Berard, Lyon
  - Centre Hospitalier Universitaire de Poitiers - Hopital la Miletrie- Pôle Régional de Cancérologie, Poitiers
  - Centre de Lutte Contre le Cancer - Institut de Cancerologie de l'Ouest - Rene Gauducheau, Saint-Herblain
  - Gustave Roussy, Villejuif
- South Korea (3):
  - Yonsei University Severance Hospital, Seoul
  - Samsung Medical Center, Seoul
  - St Mary's Hospital, The Catholic University of Korea, Seoul
- Spain (4):
  - Hospital del Mar, Barcelona
  - START Madrid-HM CIOCC Hospital Universitario HM Sanchinarro, Madrid
  - Universidad de Navarra - Clinica Universitaria de Navarra, Pamplona
  - Onkologikoa, San Sebastián
- The Royal Marsden NHS Foundation Trust - Royal Marsden Hospital, Sutton, United Kingdom